CLINICAL TRIAL: NCT01995981
Title: Individualizing Pazopanib Therapy by exploRing the Role of Early Metabolic responsE and Drug Exposure as a preDICTor for Treatment Outcome in Patients With STS
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: UMCN-ONCO-201303; 2013-003533-16 (EudraCT Number)
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2015-06

CONDITIONS: Sarcoma, Soft Tissue
Keywords: Sarcoma, Soft Tissue; Pazopanib; Positron-Emission Tomography; Pharmacokinetics; Biomarker
MeSH Terms: conditions — Sarcoma | interventions — pazopanib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced soft tissue sarcoma patients: Advanced soft tissue sarcoma patients, who have an indication for pazopanib treatment.
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib
  Other Names: Votrient

SUMMARY:
This study is a phase IV post registration prospective observational feasibility study in patients with metastatic soft tissue sarcoma. Pazopanib is the registered treatment for patients with advanced soft tissue sarcoma after chemotherapy with doxorubicin or ifosfamide.

* This study looks at the possibility of using 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG) positron emission tomography PET scans as an early biomarker of pazopanib treatment effect in patients.
* It also studies pazopanib pharmacokinetics to see if there are differences between elderly and younger patients.

The primary objectives are:

* To evaluate whether early metabolic response is correlated to clinical benefit.
* To evaluate the effect of age (≥ 70 years) on pazopanib pharmacokinetics.

The secondary objectives are:

* To evaluate whether early metabolic response (% decrease in FDG uptake due to pazopanib therapy) is correlated with pazopanib exposure.
* To evaluate whether early metabolic response (% decrease in FDG uptake due to pazopanib therapy) is correlated with the histological subtypes.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow-up.
2. Age ≥ 18 years. Patients aged 66-69 are eligible for the imaging arm of the study, however they are excluded from the assessment of altered pharmacokinetic behavior in elderly.
3. Histological confirmed diagnosis of selective subtypes of advanced soft tissue sarcoma (STS) who have received prior chemotherapy for metastatic disease or who have progressed within 12 months after (neo) adjuvant therapy. The following subtypes are eligible:

   Fibroblastic, so-called fibrohistiocytic, leiomyosarcoma, malignant glomus tumours, skeletal muscles, vascular, uncertain differentiation. The following subtypes are NOT eligible: Adipocytic sarcoma (all subtypes), all rhabdomyosarcoma that were not alveolar or pleomorphic, chondrosarcoma, osteosarcoma, Ewing tumours/primitive neuroectodermal tumor, GIST, dermatofibrosarcoma protuberance, inflammatory myofibroblastic sarcoma, malignant mesothelioma and mixed mesodermal tumours of the uterus.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. Measurable disease criteria (RECIST 1.1).
6. No radio-, chemo- or tumor specific targeted therapy within the last 4 weeks prior to study entry.
7. Adequate organ system function as defined in the research protocol.
8. Minimal evaluable lesion of ≥ 15mm.

Exclusion Criteria:

1. Prior malignancy.
2. Central nervous system (CNS) metastases at baseline, with the exception of those subjects who have previously-treated CNS metastases and who meet both of the following criteria: a) are asymptomatic and b) have no requirement for steroids or enzyme-inducing anticonvulsants in prior 6 months time interval.
3. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including.
4. Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including.
5. Corrected QT interval (QTc) > 480msecs.
6. History of any one or more of the following cardiovascular conditions within the past 6 months:

   * Cardiac angioplasty or stenting
   * Myocardial infarction
   * Unstable angina
   * Coronary artery bypass graft surgery
   * Symptomatic peripheral vascular disease
   * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
7. Poorly controlled hypertension
8. History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
9. Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer.
10. Evidence of active bleeding or bleeding diathesis.
11. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage.
12. Recent hemoptysis.
13. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
14. Unable or unwilling to discontinue use of prohibited medications listed in the research protocol for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.
15. Concurrent use of other substances known or likely to interfere with the pharmacokinetics of pazopanib
16. Treatment with any of the following anti-cancer therapies: radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of Pazopanib.
17. Administration of any non-oncologic investigational drug within 30 days or 5 half lives whichever is longer prior to receiving the first dose of study treatment.
18. Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 and/or that is progressing in severity, except alopecia.
19. For FDG-PET imaging part of the study:

    * uncontrolled diabetes mellitus
    * only evaluable tumors in brain or urinary tract, as these cannot be evaluated by FDG-PET scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced soft tissue sarcoma who have an indication for pazopanib treatment.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
FDG (18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose) uptake | baseline, 2 weeks and 8 weeks after start treatment
Pharmacokinetics (AUC) | 0, 1, 2, 3, 4, 6, 8, 10, 24 hours post-dose
  This measurement is performed at 2 weeks and 8 weeks after start treatment

SECONDARY OUTCOMES:
Adverse events (CTCAE v4.0) | 2 weeks and 8 weeks after start treatment

CONTACTS AND LOCATIONS:
Overall Officials: Winette van der Graaf, prof. PhD. MD, Principal Investigator — Radboud University Medical Center; Wim Oyen, prof. PhD. MD, Principal Investigator — Radboud University Medical Center; Nielka van Erp, PharmD. PhD., Principal Investigator — Radboud University Medical Center
Locations (2):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands
- Royal Marsden Hospital, London, United Kingdom

REFERENCES:
- [Background] van der Graaf WT, Blay JY, Chawla SP, Kim DW, Bui-Nguyen B, Casali PG, Schoffski P, Aglietta M, Staddon AP, Beppu Y, Le Cesne A, Gelderblom H, Judson IR, Araki N, Ouali M, Marreaud S, Hodge R, Dewji MR, Coens C, Demetri GD, Fletcher CD, Dei Tos AP, Hohenberger P; EORTC Soft Tissue and Bone Sarcoma Group; PALETTE study group. Pazopanib for metastatic soft-tissue sarcoma (PALETTE): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2012 May 19;379(9829):1879-86. doi: 10.1016/S0140-6736(12)60651-5. Epub 2012 May 16. PMID 22595799